CLINICAL TRIAL: NCT03367598
Title: Longitudinal Interaction Between APOA5 -1131T>C and Overweight
Brief Title: Longitudinal Interaction Between APOA5 -1131T>C and Overweight Accelerates Arterial Stiffness
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, Professor, Yonsei University
Other Study IDs: PA_fu_APOA5_rs662799
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal weight: nondiabetic and nonobese individuals (18.5 kg/m2 ≤ BMI < 25 kg/m2, n=349)
  Interventions: Genetic: rs662799 (APOA5 -1131T>C)
- Overweight: nondiabetic and nonobese individuals (25 kg/m2 ≤ BMI < 30 kg/m2, n=154)
  Interventions: Genetic: rs662799 (APOA5 -1131T>C)

INTERVENTIONS:
Genetic: rs662799 (APOA5 -1131T>C) — Among the 349 normal-weight individuals, 168 were homozygous (TT) for the T allele, 155 were heterozygous for the C allele (TC) and 26 were homozygous (CC) for the C allele of the APOA5 -1131T>C polymorphism. Among the 154 overweight individuals, 68 were homozygous (TT) for the T allele, 75 were heterozygous for the C allele (TC) and 11 were homozygous (CC) for the C allele of the APOA5 -1131T>C polymorphism.

SUMMARY:
The aim of this study is to evaluate whether the longitudinal interaction between APOA5 -1131C variants and overweight could accelerate age-related increases in arterial stiffness and circulating triglycerides in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Nondiabetic (fasting serum glucose concentration < 126 mg/dL)
* Nonobese (BMI ≥ 25 kg/m2)

Exclusion Criteria:

* Current and/or past history of cardiovascular disease
* Diabetes mellitus (fasting glucose levels ≥126 mg/dL)
* Abnormal liver or renal function
* Thyroid or pituitary disease
* Pregnancy or lactation
* Regular use of any medication

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We performed a 3-year prospective cohort study that included 800 heathy subjects (30-65 years old), of these, 503 nondiabetic and nonobese individuals were finally selected.
Sampling Method: Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Brachial-ankle PWV (baPWV) | at baseline
  cm/s
Brachial-ankle PWV (baPWV) | 3-year follow-up
  cm/s

SECONDARY OUTCOMES:
Triglyceride | at baseline
  mg/dL
Triglyceride | 3-year follow-up
  mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, PhD, Principal Investigator — Dept. of Food and Nutrition, Colleage of Human Ecology, Yonsei University